CLINICAL TRIAL: NCT05680922
Title: A First in Human Dose Escalation and Cohort Expansion Study of DLL3-directed Chimeric Antigen Receptor T-cells in Subjects With Extensive Stage Small Cell Lung Cancer
Brief Title: DLL3-Directed Chimeric Antigen Receptor T-cells in Subjects With Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Legend Biotech USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2102-1001
Record Dates: First submitted 2022-12-21; First posted 2023-01-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Large Cell Neuroendocrine Carcinoma of the Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental LB2102 (Experimental): DLL3-Directed Chimeric Antigen Receptor T-cells (CAR T)
  Interventions: Biological: LB2102

INTERVENTIONS:
Biological: LB2102 — DLL3 directed autologous Chimeric Antigen Receptor T-cells

SUMMARY:
This is a phase 1, first-in-human, open-label, multicenter, dose escalation and expansion study of DLL3-targeted chimeric antigen receptor T-cells in subjects with extensive stage small cell lung cancer or large cell neuroendocrine lung cancer.

DETAILED DESCRIPTION:
This is a phase 1, first-in-human, open-label, multicenter, dose escalation and expansion study of DLL3-targeted chimeric antigen receptor T-cells in subjects with extensive stage small cell lung cancer or large cell neuroendocrine lung cancer. The study comprises a dose-escalation component (Part A) and a cohort expansion component (Part B). Up to 41 subjects will be treated in this study. Part A will enroll and treat up to 24 subjects and Part B will be conducted after the recommended dose for expansion (RDE) has been identified in Part A and enroll up to 17 subjects. Both parts of this trial will include a Screening Period, a Pretreatment Period, a Treatment Period, a Follow-Up Period, and a Post-Progression Follow-Up Period.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and willing and able to provide a written informed consent
* Have histologically/cytologically confirmed unresectable small cell lung carcinoma (SCLC), large cell neuroendocrine lung carcinoma (LCNEC), combined SCLC, or combined LCNEC as per WHO 2021 criteria
* Subjects who have at least one prior line of standard treatment, and have progressed after or have had an insufficient response, and for whom standard treatment is intolerable, unlikely to confer significant clinical benefit, is no longer effective, or the subject declines further standard treatment
* Have available formalin-fixed, paraffin-embedded tumor specimen in a tissue block or unstained serial slides accompanied by an associated pathology report prior to enrollment. Archival or fresh biopsy tissue is required
* Presence of ≥ 1 radiologically measurable lesion per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of at least 4 months
* Have adequate organ function
* Women of childbearing potential must have a negative pregnancy test at screening using a highly sensitive serum pregnancy test (β-human chorionic gonadotropin [β-hCG])
* All subjects must agree to practice a highly effective method of contraception (failure rate of <1% per year when used consistently and correctly) from the time of signing the informed consent form (ICF) to 1 year after receiving a LB2102 infusion
* Women and men must agree not to donate eggs (ova, oocytes) or sperm, respectively, until at least 1 year after receiving a LB2102 infusion

Exclusion Criteria:

* Prior treatment with cellular immunotherapy (e.g., CAR-T) or gene therapy product
* Prior treatment with DLL3-targeted therapy
* Prior history of checkpoint inhibitor associated pneumonitis
* Clinically significant ascites, pleural or peritoneal effusions
* Known status of acquired or inherited immunodeficiency without the ability of medical control or normalization.
* Known leptomeningeal metastases
* Active or symptomatic brain metastasis. Subjects with treated brain metastasis are allowed provided definitive therapy was completed at least 2 weeks prior to enrollment with at least documented stable disease and the subject is off supraphysiologic doses of steroid for at least 7 days. Additional requirements are met per protocol.
* Active autoimmune disease receiving immunomodulatory treatments (e.g., cyclosporine or high dose systemic steroids) prior to screening as follows:

  * Within 2 weeks or 5 half-lives, whichever is longer
  * Those with steroid replacement at physiologic doses and inhaled steroids recently or currently are not excluded.
* Impaired cardiac function or clinically significant cardiac disease not controlled by medications including:
* Unstable angina or myocardial infraction within 6 months prior to apheresis.
* History of cardiomyopathy with left ventricular ejection fraction (LVEF)<45% as assessed by ECHO and MUGA scan.
* Previous or concurrent malignancy, excluding certain exceptions.
* Serious and /or uncontrolled medical condition that, in the Investigator's judgment, would cause unacceptable safety risk, interfere with study procedures or results, or compromise compliance with the protocol, such as:
* Active, uncontrolled, viral bacterial or systemic fungal infections.
* Requirement if supplemental oxygen to maintain oxygen saturation.
* Clinical evidence of dementia or altered mental status.
* Medically uncontrolled condition or insufficient recovery from an acute event within 6 months of screening.
* Subjects with known active infection with HIV, hepatitis B, and/or hepatitis C virus (HBV/HCV) are not eligible unless additional protocol requirements are met.
* subjects with HIV must be controlled on effective antiretroviral therapy for at least four weeks and have HIV viral load of less than 400 copies/mL prior to enrollment.
* subjects with active HBV must be on suppressive antiviral therapy prior to enrollment in the study.
* For subject with history of HBV and with serologic evidence of a resolved prior infection, the risk of HBV reactivation must be considered, and the need for anti-HBV prophylaxis must be carefully assessed prior to enrollment in the study.
* Subjects with untreated HCV infection may be eligible if the HCV is stable, the subject is not at risk for hepatic decompensation and the investigational cancer treatment is not expected to exacerbate the HCV infection.
* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to LB2102 excipients, such as dimethyl sulfoxide; or to fludarabine, cyclophosphamide, or tocilizumab
* Ongoing toxicity of organ functions from previous anticancer therapy that has not resolved to Grade 1 or less, except for alopecia
* Major surgery within 4 weeks prior to apheresis, or planned within 4 weeks after LB2102 administration
* Pregnant or breast-feeding
* Plans to become pregnant or breastfeed, or father a child within 1 year after receiving a LB2102 infusion
* Previous history of allogeneic hematopoietic (HSCT), organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of LB2102 and determine recommended dose for expansion (RDE) | 28 days
  Multiple doses will be tested to establish a recommended dose
To further characterize the safety and tolerability of LB2102 with the RDE identified in the dose-escalation and determine the recommended Phase 2 dose (RP2D) | 90 days
  Treatment of additional patients at the recommended dose as identified in the initial dose escalation part of the study

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of LB2102 | Through study completion, a minimum of 2 years
  Measured by Response Evaluation Criteria In Solid Tumors (RECIST)
To characterize the pharmacokinetics of LB2102 in blood | Through study completion, a minimum of 2 years
  CAR-positive T cell counts in cells/microliter (μL) blood
To evaluate the immunogenicity of LB2102 | Through study completion, a minimum of 2 years
  Number of subjects with presence of anti-LB2102 antibodies

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kentucky - Markey Cancer Center, Lexington, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No